CLINICAL TRIAL: NCT07119645
Title: A Decentralized, Randomized, Active-Controlled Clinical Trial Investigating the Effects of NT-II™ (Salmon Undenatured Type II Collagen) on Activity-Related Knee Discomfort and Functional Performance in Healthy Adults
Brief Title: NT-II™ Collagen for Joint Discomfort and Function
Acronym: NTII-JOINT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTII-HBC-001
Record Dates: First submitted 2025-06-22; First posted 2025-08-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-06

CONDITIONS: Activity-Related Knee Discomfort; Joint Discomfort; Functional Joint Pain; Functional Knee Pain; Knee Acute and Chronic Pain
Keywords: Undenatured Type II Collagen; NT-II™; Salmon Collagen; Glucosamine; Chondroitin; Joint Health; Knee Pain; Range of Motion; Activity-Related Pain; Inflammation; Decentralized Clinical Trial; Activity-related Knee Discomfort
MeSH Terms: conditions — Chronic Pain; Inflammation | interventions — Glucosamine; Chondroitin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NT-II™ 240 mg (Experimental): Participants in this arm will take one capsule of NT-II™ (Salmon Undenatured Type II Collagen) containing 240 mg daily by mouth for 12 weeks. The product is derived from enzymatically processed salmon cartilage and bone, designed to support joint health through oral tolerance mechanisms.
  Interventions: Dietary Supplement: NT-II™ (240 mg)
- NT-II™ 480 mg (Experimental): Participants in this arm will take two capsules of NT-II™ (each containing 240 mg) by mouth daily for a total daily dose of 480 mg for 12 weeks. The product is a marine-based undenatured type II collagen intended to support joint comfort and mobility.
  Interventions: Dietary Supplement: NT-II™ 480 mg
- Glucosamine/Chondroitin (Active Comparator): Participants in this arm will take a commercially available joint supplement (Kirkland) containing 1500 mg glucosamine and 1300 mg chondroitin by mouth daily for 12 weeks. This combination is commonly used to support joint structure and function and serves as the comparator in this study.
  Interventions: Dietary Supplement: Glucosamine/Chondroitin

INTERVENTIONS:
Dietary Supplement: NT-II™ (240 mg) — A once-daily capsule containing 240 mg of NT-II™, a marine-derived undenatured type II collagen supplement obtained from enzymatically processed salmon cartilage and bone. Taken orally for 12 weeks.
  Arms: NT-II™ 240 mg
Dietary Supplement: NT-II™ 480 mg — Two capsules of NT-II™ (each 240 mg), taken orally once daily for a total of 480 mg/day over 12 weeks. Sourced from salmon bone and cartilage to support joint health via oral tolerance.
  Arms: NT-II™ 480 mg
Dietary Supplement: Glucosamine/Chondroitin — A combined dietary supplement containing 1500 mg glucosamine and 1300 mg chondroitin, taken orally once daily for 12 weeks. This supplement serves as the active comparator and is widely used to support joint structure and function.
  Arms: Glucosamine/Chondroitin

SUMMARY:
The goal of this clinical trial is to learn whether a natural marine supplement called NT-II™ (Salmon Undenatured Type II Collagen) can help lower knee discomfort caused by physical activity in otherwise healthy adults. Many active people experience knee pain when performing daily movements like climbing stairs, walking long distances, or squatting, even if they do not have a medical diagnosis such as arthritis. This discomfort can limit mobility, impact exercise routines, and reduce overall quality of life. This study is being conducted to determine whether NT-II™, taken as a once-daily oral supplement, can reduce this type of activity-related knee discomfort more effectively than a commonly used joint supplement containing glucosamine and chondroitin.

The main questions the study aims to answer are:

Does NT-II™ reduce knee discomfort caused by repeated activity over a 12-week period?

Does NT-II™ improve movement and quality of life compared to glucosamine-chondroitin?

Researchers will compare two different doses of NT-II™ (240 mg and 480 mg) to glucosamine (1500 mg) plus chondroitin (1300 mg), which is used as an active comparator. All three products will be taken once daily for 12 weeks.

Participants will:

Take their assigned supplement daily by mouth for 12 weeks

Track knee discomfort once per week using a pain rating scale called a visual analog scale (VAS) while doing an activity that usually causes discomfort, such as climbing stairs, walking, or squatting

Complete short surveys online about joint function, pain, and quality of life (including KOOS and SF-12 questionnaires)

Use a mobile app to perform simple knee range of motion tests at home

Wear a fitness tracker to monitor daily physical activity, such as step count and stair climbing

Collect two small blood samples at home using a finger-prick kit to check for changes in inflammation-related biomarkers

This study is for U.S.-based adults between the ages of 20 and 65 who are in generally good health but have had mild to moderate knee discomfort caused by physical activity for at least three months. The pain must be triggered by specific weight-bearing movements and be relieved by rest. Participants must not have osteoarthritis, rheumatoid arthritis, or other joint diseases. Individuals with recent knee injuries, major surgeries, or injections in the past six months cannot take part. Participants should not be using NSAIDs, turmeric, collagen, or other joint-related supplements during the study.

All study activities will take place remotely using a secure digital platform. There are no in-person clinic visits required. Eligible participants will receive all study materials by mail, including supplements, a wearable device, and an at-home blood sample collection kit. They will also be given access to a secure digital platform (Alethios) where they can complete questionnaires, enter pain ratings, and receive study instructions. Study staff will monitor progress, check for missing data, and assist participants through secure communication tools built into the platform.

The primary outcome of the study is the change in participant-reported knee discomfort, measured using a nominated activity VAS score (VASNA), from baseline to week 12. Additional outcomes will explore changes in function, mobility, physical activity, heart rate variability, and inflammatory biomarkers. The Pain Catastrophizing Scale (PCS) will also be used to examine whether thoughts and feelings about pain influence symptom reporting and treatment response.

This trial is sponsored by Hofseth BioCare ASA and is being conducted entirely online to improve access, lower participant burden, and support real-world understanding of joint health supplements. Study results may inform the use of NT-II™ as a marine-based nutritional strategy to support joint comfort in active individuals.

DETAILED DESCRIPTION:
This is a decentralized, randomized, three-arm clinical trial evaluating the effects of NT-II™, a marine-derived undenatured type II collagen, on activity-related knee discomfort (ArKD) in otherwise healthy adults. The trial is sponsored by Hofseth BioCare ASA and conducted entirely virtually in the United States using the Alethios digital clinical trial platform.

Undenatured type II collagen has been studied for its role in promoting joint health, primarily through immune-mediated mechanisms that support oral tolerance and reduce inflammation in joint tissues. While the majority of existing evidence is based on UC-II®, derived from chicken sternum, NT-II™ offers a novel alternative derived from Norwegian Atlantic salmon (Salmo salar), embedded in a natural hydroxyapatite matrix. This study seeks to evaluate NT-II™ as a non-pharmacological intervention for individuals experiencing reproducible, activity-induced knee pain but without clinical joint disease.

Eligible participants are healthy U.S. adults aged 20 to 65, with body mass index (BMI) between 20.0 and 32.5 kg/m², who report activity-related knee discomfort of moderate intensity (VAS score 30-75 mm) for at least 3 months. Discomfort must be reliably triggered by specific knee-loading movements (e.g., stairs, squatting, walking) and relieved with rest. Individuals with clinically diagnosed osteoarthritis or recent joint injury are excluded.

Following screening and a one-week run-in period (with symptom tracking only), participants are randomized in a 1:1:1 ratio to receive one of three interventions for 12 weeks:

NT-II™ standard dose - 240 mg/day

NT-II™ high dose - 480 mg/day

Glucosamine (1500 mg) + Chondroitin (1300 mg) - active comparator

The primary endpoint is the change in self-reported knee discomfort on a participant-nominated visual analog scale (VASNA) - an activity-specific VAS ranging from 0 to 100 mm - from baseline to week 12. Participants nominate their most aggravating activity (e.g., stair descent), and VAS pain scores are collected weekly throughout the trial.

Secondary outcomes include:

Subscale scores from the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire

Range of motion assessments (via the validated Curovate app)

Health-related quality of life (SF-12)

Daily activity metrics (e.g., step count, floors climbed) via wearable devices

Heart rate variability (HRV) recovery time as a biomarker of physiological resilience

Pain Catastrophizing Scale (PCS) to assess psychological contributors to pain reporting

The study is open-label, with centralized, blinded data analysis for biomarkers and PROMs. Outcome data are collected entirely remotely via the Alethios platform, wearable devices, mobile apps, and at-home blood collection kits.

This trial will assess both dose-response effects of NT-II™ and its comparative effectiveness versus glucosamine-chondroitin. It is designed to generate high-quality clinical evidence for NT-II™ in a functional knee discomfort population, while also exploring digital trial infrastructure, decentralized methodologies, and personalized symptom reporting frameworks. By integrating subjective and objective metrics, the study aims to enhance understanding of nutritional joint interventions in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 65 years.
* Self-reported, reproducible knee discomfort associated with any knee-loading activities for at least 3 months prior to screening.
* Discomfort must occur in at least one knee during a nominated aggravating activity at least twice per week and subside with rest.
* VAS rating of 30 mm to 75 mm during the past week for the nominated activity.
* No current diagnosis of structural joint disease (e.g., osteoarthritis).
* Engages in physical activity involving knee-loading movements at least twice weekly for 20+ minutes.
* BMI between 20.0 and 32.5 kg/m².
* In good general health with no significant medical comorbidities.
* Able and willing to provide informed consent.
* Capable of completing study procedures remotely using mobile technology.

Exclusion Criteria:

* Persistent knee pain at rest or recent acute lower-limb trauma.
* Diagnosed structural or inflammatory joint disorders.
* Current or recent physiotherapy targeting knee pain (within 6 months).
* Allergy to fish or any study product ingredients.
* Scheduled lower-limb surgery during the study period.
* Other musculoskeletal disorders affecting ambulation.
* Recent joint injections (within 3 months).
* Use of joint supplements in the past 3 months.
* Use of analgesics ≥3 days/week in the past 3 months.
* NSAIDs/acetaminophen use is permitted with restrictions:
* Not within 24 hours of blood sampling or VAS assessments.
* Must be documented.
* Chronic use of medications that affect musculoskeletal symptoms (e.g., muscle relaxants, gabapentinoids) unless infrequent (≤2x/week) and not within 24 hours of assessments.
* Regular use of PPIs (>3x/week in past month).
* Systemic corticosteroids, immunosuppressants, or opioids within 4 weeks.
* Unstable weight or significant recent dietary changes.
* Significant medical conditions (e.g., cancer, hepatic/renal impairment, CVD, thyroid disease, diabetes).
* Neurological, cognitive, or psychiatric disorders affecting participation.
* Use of tobacco/nicotine or other substances.
* Diagnosed sleep disorders.
* Strict vegan diet or sedentary lifestyle.
* Inability to swallow capsules.
* Pregnant, breastfeeding, or planning pregnancy.
* Women of childbearing potential not using contraception.
* Participation in another interventional clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-19 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in participant-nominated activity-related knee discomfort (VASNA for pain) from baseline to week 12 | Baseline to Week 12
  Each participant will identify a specific weight-bearing activity (e.g., stair descent, walking, or squatting) that consistently causes knee discomfort. Pain intensity will be rated on a 100 mm visual analog scale (VAS) for that activity at baseline and again at week 12. The primary outcome is the change in VASNA score from baseline to week 12.

SECONDARY OUTCOMES:
Longitudinal Change in Nominated VAS | Baseline through Week 12.
  Participants will rate knee discomfort weekly using a 100 mm visual analog scale (VAS) for their nominated aggravating activity. Mixed-effects models will assess changes over time and treatment group-by-time interactions, including linear and nonlinear patterns.
Cumulative symptom improvement assessed by Incremental Area Under the Curve (iAUC) of weekly Nominated VAS | Baseline to Week 12
  The incremental area under the curve (iAUC) will be calculated for weekly Nominated VAS scores from baseline to Week 12 to evaluate cumulative symptom improvement across all treatment arms.
KOOS Subscale Changes | Baseline to Week 6 and Week 12
  Change from baseline to Week 6 and Week 12 in subscale scores from the Knee Injury and Osteoarthritis Outcome Score (KOOS), including Pain (9 items), Symptoms (7 items), Activities of Daily Living (17 items), Sport and Recreation Function (5 items), and Knee-related Quality of Life (4 items). Each item is rated using a 5-point Likert scale, from 0 ("No problems") to 4 ("Extreme problems"). Subscale scores are calculated as the sum of item scores, then transformed to a 0-100 scale, where 0 represents extreme knee problems and 100 represents no problems. Subscales are analyzed separately to evaluate domain-specific effects across treatment arms.
KOOS Item-Level Functional Response | Baseline to Week 6 and Week 12
  Change from baseline to Week 6 and Week 12 in selected item-level responses from the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire. Items reflect functional aspects of pain, symptoms, and mobility, including: Pain (Items 1, 4, 9), Symptoms (Items 2, 3, 7), Activities of Daily Living (Items 1, 4, 9, 10), Sport and Recreation Function (Items 3, 4), and Quality of Life (Items 1-4). Each item is rated using a 5-point Likert scale from 0 ("No problems") to 4 ("Extreme problems"), with scores transformed to a 0-100 scale where higher scores indicate better outcomes. Between-group differences in activity-specific pain and function patterns will be explored to assess targeted effects of treatment.
SF-12 Health Survey Score Changes | Baseline to Week 12
  Change in scores from the 12-Item Short Form Health Survey (SF-12) from baseline to Week 12 will be compared across treatment arms. The SF-12 generates two composite summary scores-Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12)-each scaled from 0 to 100, where higher scores indicate better health status, including physical, mental, and social functioning. The SF-12 is an abbreviated version of the SF-36 and reliably reproduces its summary scores with less participant burden. Changes in PCS-12 and MCS-12 will be evaluated to assess improvements in quality of life associated with each intervention.
Validated Mobile Application Self-Assessed Knee Range of Motion | Baseline to Week 12
  Self-reported, app-guided measurements of knee flexion and extension ROM using the Curovate mobile app will be compared from baseline to Week 12 across intervention groups.
Participant-Reported Satisfaction With Treatment and Study Experience | Week 12
  At Week 12, participants will rate their overall satisfaction with the treatment and study experience using a global self-assessment and an optional free-text comment. Satisfaction responses will be categorized as positive, neutral, or negative, based on participant selection or the sentiment of free-text responses. Coded values will be assigned as follows: positive = 1, neutral = 0, negative = -1. Categorized satisfaction scores will be compared across treatment arms to explore differences in perceived benefit and study experience.
  Unit of Measure: Categorized satisfaction score derived from participant responses (coded as -1 = negative, 0 = neutral, 1 = positive; higher scores indicate greater satisfaction)
Heart Rate Variability (HRV) | Baseline through week 12 (continuous)
  Wearable-derived heart rate variability (HRV) will be measured to assess physiological stress response as a proxy for chronic autonomic sympathetic/parasympathetic tone.
Exploratory Analysis of Pain Catastrophizing and Its Influence on Pain Perception | Baseline to Week 12
  To assess the influence of cognitive-affective factors on pain perception, changes in VAS Nominated Activity-related Pain (VASNA) and KOOS subscale scores will be analyzed stratified by baseline Pain Catastrophizing Scale (PCS) scores (e.g., low vs. high). This exploratory analysis aims to determine whether baseline catastrophizing affects perceived symptom severity and response to intervention.
  Unit of Measure for VASNA: VAS score (0-100; higher scores indicate greater pain) Unit of Measure for KOOS subscales: KOOS subscale score (0-100; higher scores indicate better outcomes)
Change in Mean Daily Step Count Measured by Smartwatch | Baseline through Week 12 (continuous)
  Mean daily step count, recorded continuously by smartwatch, will be calculated from baseline through Week 12. Changes in step count will be assessed across treatment arms to evaluate differences in overall physical activity levels.
  Unit of Measure: Steps per day
Change in Mean Daily Floors Climbed Measured by Smartwatch | Baseline through Week 12 (continuous)
  Mean daily number of floors climbed, recorded by smartwatch using barometric and motion sensors, will be measured continuously from baseline through Week 12. Changes in floors climbed will be analyzed between groups to assess changes in vertical mobility and lower-body functional activity.
  Unit of Measure: Floors per day.

OTHER OUTCOMES:
Smartwatch-Derived Sleep Quality Score (Exploratory) | Baseline through weeks 12 (continuous)
  Sleep quality will be assessed using composite scores derived from smartwatch data, including metrics such as total sleep time, sleep efficiency, and time in different sleep stages (e.g., deep, light, REM). A standardized sleep quality index will be calculated and compared between participants receiving NT-II™ (any dose) and those receiving glucosamine-chondroitin.
  Unit of Measure: Composite sleep quality score (0-100; higher scores indicate better sleep quality)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the proprietary nature of the intervention, data privacy considerations related to remote monitoring technologies, and the absence of a pre-specified data sharing agreement. The sponsor may consider future data sharing requests on a case-by-case basis in accordance with applicable privacy regulations and scientific relevance.